CLINICAL TRIAL: NCT05490992
Title: In-person and Telehealth Versions of Behavioral Skills Training to Reduce Car Seat Misuse
Brief Title: Behavioral Skills Training Methods to Reduce Car Seat Misuse
Acronym: BSTCPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro Consumer Safety - Public Health Behavior Solutions (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, James DeCarli, Injury & Neuroepidemiologist, Pro Consumer Safety - Public Health Behavior Solutions
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BSTCPS2022
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Motor Vehicle Injury
Keywords: motor vehicle occupant injury; car seat misuse; car seat education; Behavioral Skills Training; Telehealth

STUDY DESIGN:
Intervention Model Description: This study is a quasi-experimental within-subjects group design. It consists of two experiments that included an equal number of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Car seat check-up traditional car seat educational method (No Intervention): Experiment-1a: This included 600 expectant parents who were educated by a certified child passenger safety technician with a traditional car seat educational approach. All participants were assessed at baseline, no-intervention traditional education, and follow-up, between June 1, 2015 and May 30, 2016
- Behavioral Skills Training In-person Group A (Experimental): Experiment-1b: This included another 600 expectant parents who were educated by a certified child passenger safety technician an in-person Behavioral Skills Training (BST) approach. All participants were assessed at baseline, BST, and follow-up, between June 1, 2016 and May 30, 2017.
  Interventions: Other: Behavioral Skills Training In-person
- Behavioral Skills Training In-person Group B (Experimental): Experiment-2a: This included another 600 expectant parents who were educated by a certified child passenger safety technician an in-person Behavioral Skills Training (BST) approach. All participants were assessed at baseline, BST, and follow-up, between June 1, 2018 and June 30, 2019.
  Interventions: Other: Behavioral Skills Training In-person
- Behavioral Skills Training Telehealth (Experimental): Experiment-2b: This included another 600 expectant parents who were educated by a certified child passenger safety technician a virtual telehealth version of Behavioral Skills Training (BST). All participants were assessed at baseline, BST-Telehealth, and follow-up, between April 1, 2020 and December 31, 2021.
  Interventions: Other: Behavioral Skills Training In-person

INTERVENTIONS:
Other: Behavioral Skills Training In-person — Both an in-person and virtual telehealth version of Behavioral Skills Training (BST) was compared to the "Car seat check-up traditional car seat educational method" and BST telehealth was compared to BST in-person.
  Other Names: Behavioral Skills Training Telehealth
  Arms: Behavioral Skills Training In-person Group A; Behavioral Skills Training In-person Group B; Behavioral Skills Training Telehealth

SUMMARY:
The purpose of this study is to assess the effectiveness of child passenger educational methods to measure their ability to effectively reduce car seat misuse. The study will assess the traditional child passenger educational method delivered by a child passenger safety technician by comparing it to an in-person and virtual telehealth Behavioral Skills Training approach to reduce car seat misuse.

DETAILED DESCRIPTION:
This study of 2,449 expectant couples involved two experiments. Experiment-1: included 1,224 participants, comparing 600 participants receiving no intervention and 600 participants receiving education with behavioral skills training (BST) in-person.

Experiment-2: included 1,224 participants, comparing 600 participants receiving BST-in-person to BST with telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 7-month gestation and their partner, living within Los Angeles, Ventura, Orange, San Bernardino or Riverside counties; consented to the study and follow-up evaluation; and at the time of session had their child restraint system(s) and vehicle(s) available.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2448 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
child restraint misuse | 12 months
  Incidence of misuse

CONTACTS AND LOCATIONS:
Overall Officials: James M DeCarli, PhD, MPH, Principal Investigator — Public Health Behavior Solutions/State of California
Locations (1):
- Pro Consumer Safety/Pro Car Seat Safety - NHTSA CPS Inspection Station, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boutain AR, Sheldon JB, Sherman JA. Evaluation of a telehealth parent training program in teaching self-care skills to children with autism. J Appl Behav Anal. 2020 Jul;53(3):1259-1275. doi: 10.1002/jaba.743. Epub 2020 Jul 13. PMID 32657441
- [Result] Carnett A, Hansen S, Tullis C, Machalicek W. Using behavioural skills training via telehealth to increase teachers use of communication interventions and increase student use of speech-generating devices in a high school functional skills classroom. J Intellect Disabil Res. 2021 Feb;65(2):133-148. doi: 10.1111/jir.12794. Epub 2020 Nov 13. PMID 33185000
- [Result] Dickson MJ, Vargo KK. Training kindergarten students lockdown drill procedures using behavioral skills training. J Appl Behav Anal. 2017 Apr;50(2):407-412. doi: 10.1002/jaba.369. Epub 2017 Jan 11. PMID 28078673
- [Result] Edgemon AK, Rapp JT, Brogan KM, Richling SM, Hamrick SA, Peters RJ, O'Rourke SA. Behavioral skills training to increase interview skills of adolescent males in a juvenile residential treatment facility. J Appl Behav Anal. 2020 Sep;53(4):2303-2318. doi: 10.1002/jaba.707. Epub 2020 Apr 17. PMID 32301517
- [Result] Executive Order. No. N-33-20 H.S.C. § 8567 8627 8665, 2020. https://covid19.ca.gov/img/Executive-Order-N-33-20.pdf
- [Result] Giannakakos AR, Vladescu JC, Simon R. Teaching installation and use of child passenger safety restraints. J Appl Behav Anal. 2018 Oct;51(4):915-923. doi: 10.1002/jaba.493. Epub 2018 Jul 13. PMID 30006981
- [Result] Himle MB, Wright KA. Behavioral skills training to improve installation and use of child passenger safety restraints. J Appl Behav Anal. 2014 Fall;47(3):549-59. doi: 10.1002/jaba.143. Epub 2014 Jun 3. PMID 24891092
- [Result] Hoffman BD, Gallardo AR, Carlson KF. Unsafe from the Start: Serious Misuse of Car Safety Seats at Newborn Discharge. J Pediatr. 2016 Apr;171:48-54. doi: 10.1016/j.jpeds.2015.11.047. Epub 2015 Dec 18. PMID 26707620
- [Result] Miltenberger, Raymond G. "Behavioral Skills Training Procedures." (2016) Behavior Modification Principles and Procedures, 6th ed., Cenage Learning, pp. 223-242.
- [Result] National Center for Statistics and Analysis. (2022, March - revised). Children: 2019 data. (Traffic Safety Facts. Report No. DOT HS 813 122). National Highway Traffic Safety Administration
- [Result] National Highway Traffic Safety Administration. (2004, January). Misuse of Child Restraints (DOT HS 809 671). United States, Department of Transportation. https://www.nhtsa.gov/sites/nhtsa.gov/files/documents/809671.pdf
- [Result] National Highway Traffic Safety Administration. (2022). The Right Seat. Parents Central-From Car Seats To Car Keys: Keeping Children Safe. Retrieved July 24, 2022, from https://one.nhtsa.gov/links/ParentsCentral/CarSeats.htm#.
- [Result] Raymond, P. (2018, July). Additional Analysis of National Child Restraint Use Special Study: Child Restraint Misuse (DOT HS 812 527). Traffic Safety Facts: Research note. https://www.nhtsa.gov/sites/nhtsa.gov/files/documents/13648-additional_analysis_of_ncruss_071718_v3_tag.pdf
- [Result] Rios, D., Schenk, Y. A., Eldridge, R. R., & Peterson, S. M. (2020). The Effects of Remote Behavioral Skills Training on Conducting Functional Analyses. Journal of Behavioral Education, 29(2), 449-468. https://doi.org/10.1007/s10864-020-09385-3.
- [Result] Shigekawa E, Fix M, Corbett G, Roby DH, Coffman J. The Current State Of Telehealth Evidence: A Rapid Review. Health Aff (Millwood). 2018 Dec;37(12):1975-1982. doi: 10.1377/hlthaff.2018.05132. PMID 30633674
- [Result] Sump LA, Richman DM, Schaefer AM, Grubb LM, Brewer AT. Telehealth and in-person training outcomes for novice discrete trial training therapists. J Appl Behav Anal. 2018 Jul;51(3):466-481. doi: 10.1002/jaba.461. Epub 2018 Apr 23. PMID 29683185
- [Result] Thomas BR, Lafasakis M, Spector V. Brief Report: Using Behavioral Skills Training to Teach Skateboarding Skills to a Child with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Dec;46(12):3824-3829. doi: 10.1007/s10803-016-2900-8. PMID 27632185
- [Result] Wegner MV, Girasek DC. How readable are child safety seat installation instructions? Pediatrics. 2003 Mar;111(3):588-91. doi: 10.1542/peds.111.3.588. PMID 12612241
- [Result] Wijesooriya NR, Mishra V, Brand PLP, Rubin BK. COVID-19 and telehealth, education, and research adaptations. Paediatr Respir Rev. 2020 Sep;35:38-42. doi: 10.1016/j.prrv.2020.06.009. Epub 2020 Jun 18. PMID 32653468
- [Result] WISQARS (Web-Based Injury Statistics Query and Reporting System) Injury Center CDC. Centers for Disease Control and Prevention, Centers for Disease Control and Prevention, 1 July 2020, www.cdc.gov/injury/wisqars/index.html.